CLINICAL TRIAL: NCT00822991
Title: Sonazoid Enhanced Liver Cancer Trial for Early Detection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kindai University (Other)
Responsible Party: Japan Liver Oncology Group, Kinki University School of Medicine, Gastroenterology and Hepatology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: JLOG08001; UMIN000001612
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2009-01

CONDITIONS: Hepatocellular Carcinoma; Liver Cirrhosis; Hepatitis B; Hepatitis C
Keywords: Sonazoid; Early detection; Hepatocellular carcinoma; Liver cirrhosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis; Hepatitis B; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group of CE-US (Active Comparator): screening by CE-US using Sonazoid(TM) in the postvascular phase every 3-5 months
  Interventions: Device: CE-US (Sonazoid™)
- Group of B-mode US (Active Comparator): screening by conventional B-mode US every 3-5 months
  Interventions: Device: B-mode US

INTERVENTIONS:
Device: CE-US (Sonazoid™) — screening by CE-US using Sonazoid(TM) in the postvascular phase every 3-5 months
  Other Names: Sonazoid Group
  Arms: Group of CE-US
Device: B-mode US — screening by conventional B-mode US every 3-5 months
  Other Names: B-mode Group
  Arms: Group of B-mode US

SUMMARY:
The aim of this study is to prove usefulness of contrast-enhanced ultrasound (CE-US) using Sonazoid (TM) in the early detection of HCC as compared with conventional B-mode ultrasound (B-mode US) for hepatitis virus related cirrhosis, who are defined as super high-risk patients for hepatocarcinogenesis,Furthermore, to analyze whether early detection of HCC by CE-US has a survival benefit than that by B-mode US.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 20
2. HBV or HCV related liver cirrhosis
3. No history of HCC
4. Diagnosed as liver cirrhosis histologically or clinically Histologically confirmed by liver biopsy Confirmed by formula of diagnosing cirrhosis Radiological finding Finding of portal hypertension Platelet<130,000
5. Inpatient or outpatient
6. Patients who signed a written informed consent form

Exclusion Criteria:

1. History of hypersensitivity to egg yolk
2. Pregnant or lactating women and women who may be pregnant
3. Severe liver dysfunction(AST, ALT,or BIL level >10ULN
4. Associated with HCC
5. Patients receiving interferon
6. Age under 20
7. Judged by investigator not to be appropriate for inclusion in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2009-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Size of HCC which is detected first | 10 years

SECONDARY OUTCOMES:
Time to detection of HCC | 10 years
The improvement of prognosis of patients who are diagnosed in this study | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Masatoshi Kudo, professor, Principal Investigator — Kindai University
Locations (1):
- Kinki University School of Medicine, Department of Gastroenterology and Hepatology, Ōsaka-sayama, Osaka, Japan

REFERENCES:
- [Derived] Kudo M, Hatanaka K, Kumada T, Toyoda H, Tada T. Double-contrast ultrasound: a novel surveillance tool for hepatocellular carcinoma. Am J Gastroenterol. 2011 Feb;106(2):368-70. doi: 10.1038/ajg.2010.432. No abstract available. PMID 21301463